CLINICAL TRIAL: NCT00743756
Title: Study of a Home Delivered Meal Program on Obese Elderly African American Subjects With T2Dm
Brief Title: Study of a Home Delivered Meal Program on Obese Elderly African American Subjects With Type 2 Diabetes Mellitus (DM)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow patient enrollment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1404-2005
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Obesity; Diabetes
Keywords: obesity; diabetes; endothelial function; insulin sensitivity
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): A total of 20 African-American patients with type 2 diabetes will be randomized to receive home-delivered meals for twelve consecutive months. In addition, the subjects received diabetes education at every visit (8 clinic visits and 8 phone calls)
  Interventions: Dietary Supplement: home-delivered meals
- 2 (Experimental): A total of 20 African-American patients with type 2 diabetes will be randomized to receive home-delivered meals for six consecutive months. In addition, the subjects received diabetes education for up to twelve months(8 clinic visits and 8 phone calls)
  Interventions: Dietary Supplement: home-delivered meals
- 3 (Other): 20 subjects received 12 months of diabetes education (8 clinic visits and 8 phone calls)
  Interventions: Behavioral: diabetes education for 12 months

INTERVENTIONS:
Dietary Supplement: home-delivered meals — 3 diabetic meals per day, 7 days per week for 12 months
  Arms: 1
Dietary Supplement: home-delivered meals — diabetic meals 3 times per day, 7 days a week for six months
  Arms: 2
Behavioral: diabetes education for 12 months — subjects in this group received diabetes education for 12 months
  Arms: 3

SUMMARY:
The purpose of this study is to assess the impact of home-delivered Medical Nutrition Therapy on clinical outcomes for persons with diabetes. The primary outcomes of this studies include A1c (A1C), blood glucose, blood pressure, Body Mass Index, lipid levels and other measures of disease progression and management as well as costs of medical care provided throughout the intervention period.

DETAILED DESCRIPTION:
Data collected as a result of this project will be evaluated in aggregate to demonstrate the potential impacts on health and medical costs available through this type of intervention, with long-term goals of reducing disability and deaths due to chronic disease.

ELIGIBILITY:
Inclusion Criteria:

1. African-American subjects
2. Males or females 65 - 85 years of age
3. Body mass index (BMI) equal to or greater than 30 kg/m2
4. Fasting blood glucose less than 300 mg/dL and HbA1c less than 9.0%
5. Ability to understand and be willing to adhere to the study protocol
6. A known history of type 2 diabetes mellitus greater than 3 months, receiving either diet alone or oral antidiabetic agents (sulfonylureas, metformin, thiazolidinediones).

Exclusion Criteria:

1. Subjects with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state.
2. Patients with clinically relevant hepatic disease or impaired renal function, as shown by a serum creatinine greater than 3.0 mg/dL.
3. Mental condition rendering the subject unable to understand the scope of the study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-04; Primary Completion 2009-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Weight Loss in the elderly african american population | 6 months to 1 year

SECONDARY OUTCOMES:
Endothelial Function (assessed by pulse-wave analysis); sympathetic activity; insulin sensitivity | 6 months to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo E Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States